CLINICAL TRIAL: NCT05844189
Title: Physiotherapy Treatment With Capacitive Resistive Monopolar Radiofrecuency in Young Women With Dyspareunia
Acronym: [CRMRF]
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escoles Universitaries Gimbernat (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EUGimbernat
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Dyspareunia; Female
Keywords: Capacitive Resistive Monopolar Radiofrecuency; Sexual Dysfunction, Physiological; Pelvic floor; Physical Therapy Modalities; Musculoskeletal Manipulations
MeSH Terms: conditions — Dyspareunia; Sexual Dysfunction, Physiological | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): CRMRF and physical therapy modalities on pelvic floor.
  Interventions: Procedure: Physical therapy modalities on pelvic floor (manual therapy); Device: CRMRF
- Sham Group (Sham Comparator): Only physical therapy modalities on pelvic floor. In this Arm the CRMRF is off.
  Interventions: Procedure: Physical therapy modalities on pelvic floor (manual therapy); Device: Sham CRMRF

INTERVENTIONS:
Procedure: Physical therapy modalities on pelvic floor (manual therapy) — Intravaginal treatment (perineal massage)
Device: CRMRF — CRMRF application on pelvic floor:
  * Externally over the urogenital triangle of the patient,
  * Intracavitary application (intravaginal)
  * Externally over the urogenital triangle of the patient while the physical therapist performs the intracavitary manual therapy (intravaginal),
  The device used is named "Intradermik" and it is the portable CRMRF device of the brand RÖS'S Estética SL.
  It has these features:
  * Frequency: 448kHz
  * Capacitive power: 450 voltamperes
  * Resistive power: 200 watts
  Arms: Treatment Group
Device: Sham CRMRF — The physical therapist applies the same treatment as the Treatment Group but the device is switched off.
  Arms: Sham Group

SUMMARY:
The hypothesis of this study is that capacitive-resistive monopolar radiofrecuency (CRMRF) with vaginal manual physiotherapy improves sexual health in young women suffering from dyspareunia (pain during sexual intercourse). The realization of studies that help to know the therapeutic possibilities in the field of dyspareunia seems necessary, taking into account the number of women affected, as well as the deficits of scientific evidence in this field.

The main objective of this study is to analyze whether the use of CRMRF brings additional benefits to the results of manual therapy on dyspareunia in young women.

Likewise, it intends to analyze the data for two secondary objectives:

1. Analyze changes in different areas of women's sexual function in young people with dyspareunia through treatment (Desire, arousal, lubrication, orgasm, satisfaction and pain).
2. Study if the use of CRMRF is an added benefit in personal perception while receiving treatment.

DETAILED DESCRIPTION:
After being informed of the study objectives, inclusion and exclusion criteria, and study methodology, all patients have signed informed consents. The participation of women in this study is entirely voluntary and if, during the course of the study, a participant decides to withdraw, she can do it freely at the time she considers appropriate, without the need to give explanations.

At week 0, patients who meet the eligibility requirements will be randomized using "Random.org" in a single-blind manner (participant) in two Arms:

1. Treatment Group (CRMRF and physical therapy modalities on pelvic floor)
2. Sham Group (only physical therapy modalities on pelvic floor).

There will be 4 identical treatment sessions (one each week). These sessions are protocolized. Data collection will be carried out before the first session, after the last session and 12 weeks after the end of the treatment. The approximate duration of each session is 40 minutes. Sessions with data collection will be approximately between 45 minutes to 1 hour.

During the first visit, patients will be asked to answer a series of questions and respond to some questionnaires (FSFI, Female Sexual Function Index and FSM, Women's Sexual Function). The results of the different tests carried out, as well as all the documentation referring to the participants, are totally confidential and will only be available to the main researcher, the collaborators and the health authorities competent, if applicable.

All necessary security measures so that study participants are not identified and confidentiality measures in all cases will be complete, in accordance with Regulation 2016/679 of the European Parliament and of the Council of April 27, 2016 on the + protection of natural persons (RGPD) and Organic Law 3/2018, of December 5, Protection of Personal Data and Guarantee of Digital Rights (LOPD-GDD).

During treatment, the patient will be placed in the supine position for the treatment, in litotonic position, because in this position the abdominal muscles and coxofemoral joints will be relaxed. The manual therapy techniques in the two groups will be based on Thiele's perineal massage, which consists of a massage from the origin to the insertion of the levator anus muscle with an amount of pressure tolerable by the patient. The maneuver will be performed by performing a back and forth movement over the entire palpable surface of muscle.

CRMRF will be performed on the treatment group with two types of active electrodes that, throughout the treatment, will be kept moving to avoid heat concentration.

1. An external capacitive electrode, flat, stainless steel and coated with polyamide of 3cm diameter (ECE), which will act on the superficial tissues, skin, mucosa and muscle. It will be used externally bordering the external vaginal lips while the physiotherapist performs the perineal massage with the other hand.
2. An internal, cylindrical, stainless steel resistive electrode, 8 cm long and 1.5 cm in diameter (ERI). It has a plastic screw-on cap to prevent heat concentration. The application will be endocavitary, in direct contact with the intravaginal tissue of the woman.

Throughout all the treatment the patient will have a passive electrode on her back, which will be a rectangular return plate. To perform the treatment, an Intradermik equipment (Rös's Estética), a conductive gel (Clear Ultrasound Gel, OXD Professional Care, REF US-C1) and the 2 different types of electrodes are used.

Participants will be blinded. As a masking technique, patients will be told that the intervention can produce a sensation of increased temperature in the area of application but that it does not always have to occur. Placing of the device will not allow participants to see the monitor. In the Sham Group, the CRMRF device is off.

The data obtained as study variables will be coded during the study, processed and analyzed.The sample population to be used in the analyses will include all participants who meet all inclusion criteria, except those who have decided to leave the study before its completion.

Statistical analysis will be performed with IBM SPSS Statistics (v20) software to assess the primary and secondary objectives and hypotheses of the study, including:

* Tests of normality of the variables.
* Analysis of the description variables of the complete sample: percentages, contingency tables, descriptive statistics (mean, standard deviation, median, minimum and maximum).
* Analysis of the sample description variables, by groups: percentages, contingency tables, descriptive statistics (mean, standard deviation, median, minimum and maximum).
* Comparison of means in related samples, separated by groups: T-test for mean difference (variables with normal distribution) and non-parametric Wilcoxon test (variables with non-normal distribution). The following comparisons are made: Final - Initial, ReTest - Final, ReTest - Initial.
* Comparison of means between groups.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 30 years old.
* Women who have pain during sexual intercourse, classified as dyspareunia superficial in the last 12 months.

Exclusion Criteria:

* Use of antidepressants.
* Pregnancy and lactation.
* Cardiac pathologies.
* Epilepsy.
* Acute inflammatory process.
* Pacemaker.
* Skin or mucous infections in the urogenital area.
* Any alteration that prevents the understanding of the informed consent.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-02-09 (Actual)

PRIMARY OUTCOMES:
Pain in sexual intercourse | Five months
  The pain was described using the anamnesis, the pain score of the "FSFI" scale (Female Sexual Function Index) and the scale of pain "VAS" (Visual Analogue Scale) that is a numerical rating scale that goes from zero to ten. Zero represents the absence of pain and ten the greatest pain that the patient can imagine.
  The pain was described also using vaginal dilators and seeing at which measure the pain begins.

SECONDARY OUTCOMES:
Female sexual function | Five months
  The female sexual function was described using the "FSFI" (Female Sexual Function Index) and the "FSM" (Women's Sexual Function).
Quality of sexual relations | Five months
  The quality of sexual relations was described using the scale "VAS" (Visual Analogue Scale) that is a numerical rating scale that goes from zero to ten. Zero represents the absence of quality of sexual relations and ten the best quality of sexual relations that the patient can imagine, the score of satisfaction of the "FSFI" (Female Sexual Function Index) and the score of "FSM" (Women's Sexual Function).
Problems with vaginal penetration | Five months
  The problems with vaginal penetration were described using the scale "FSM" (Women's Sexual Function).
State of the musculature of the pelvic floor | Five months
  The state of the musculature of the pelvic floor was described using the physical exploration of the patient and a device called "EPI-No" that can detect pain by stretching.
Perception of treatment | Five months
  The perception of treatment was described using specific questions in the anamnesis.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Abelló Pla, MSc, Principal Investigator — Escoles Universitaries Gimbernat; Jordi Esquirol Caussa, PhD, Study Director — Escoles Universitaries Gimbernat; Judit Lleberia, Study Director — Universitat Autònoma de Barcelona
Locations (1):
- Escoles Universitaries Gimbernat, Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Thomten J. Living with genital pain: Sexual function, satisfaction, and help-seeking among women living in Sweden. Scand J Pain. 2014 Jan 1;5(1):19-25. doi: 10.1016/j.sjpain.2013.10.002. PMID 29913665
- [Result] Elmerstig E, Wijma B, Swahnberg K. Young Swedish women's experience of pain and discomfort during sexual intercourse. Acta Obstet Gynecol Scand. 2009;88(1):98-103. doi: 10.1080/00016340802620999. PMID 19140047
- [Result] Hendrickx L, Gijs L, Enzlin P. Age-related prevalence rates of sexual difficulties, sexual dysfunctions, and sexual distress in heterosexual women: results from an online survey in flanders. J Sex Med. 2015 Feb;12(2):424-35. doi: 10.1111/jsm.12725. Epub 2014 Oct 27. PMID 25345486
- [Result] Mitchell KR, Geary R, Graham CA, Datta J, Wellings K, Sonnenberg P, Field N, Nunns D, Bancroft J, Jones KG, Johnson AM, Mercer CH. Painful sex (dyspareunia) in women: prevalence and associated factors in a British population probability survey. BJOG. 2017 Oct;124(11):1689-1697. doi: 10.1111/1471-0528.14518. Epub 2017 Jan 25. PMID 28120373
- [Result] Demirel G, Golbasi Z. Effect of perineal massage on the rate of episiotomy and perineal tearing. Int J Gynaecol Obstet. 2015 Nov;131(2):183-6. doi: 10.1016/j.ijgo.2015.04.048. Epub 2015 Jul 26. PMID 26410801
- [Result] Leon-Larios F, Corrales-Gutierrez I, Casado-Mejia R, Suarez-Serrano C. Influence of a pelvic floor training programme to prevent perineal trauma: A quasi-randomised controlled trial. Midwifery. 2017 Jul;50:72-77. doi: 10.1016/j.midw.2017.03.015. Epub 2017 Mar 27. PMID 28391147
- [Result] Takeuchi S, Horiuchi S. Randomised controlled trial using smartphone website vs leaflet to support antenatal perineal massage practice for pregnant women. Women Birth. 2016 Oct;29(5):430-435. doi: 10.1016/j.wombi.2016.01.010. Epub 2016 Feb 19. PMID 26906970
- [Result] Spottorno J, Gonzalez de Vega C, Buenaventura M, Hernando A. Influence of electrodes on the 448 kHz electric currents created by radiofrequency: A finite element study. Electromagn Biol Med. 2017;36(3):306-314. doi: 10.1080/15368378.2017.1354015. Epub 2017 Jul 31. PMID 28759286
- [Result] Silva AP, Montenegro ML, Gurian MB, Mitidieri AM, Lara LA, Poli-Neto OB, Rosa E Silva JC. Perineal Massage Improves the Dyspareunia Caused by Tenderness of the Pelvic Floor Muscles. Rev Bras Ginecol Obstet. 2017 Jan;39(1):26-30. doi: 10.1055/s-0036-1597651. Epub 2016 Dec 27. PMID 28027568
- [Result] Kumaran B, Watson T. Thermal build-up, decay and retention responses to local therapeutic application of 448 kHz capacitive resistive monopolar radiofrequency: A prospective randomised crossover study in healthy adults. Int J Hyperthermia. 2015;31(8):883-95. doi: 10.3109/02656736.2015.1092172. Epub 2015 Nov 2. PMID 26524223
- [Result] Trahan J, Leger E, Allen M, Koebele R, Yoffe MB, Simon C, Alappattu M, Figuers C. The Efficacy of Manual Therapy for Treatment of Dyspareunia in Females: A Systematic Review. J Womens Health Phys Therap. 2019 Jan-Mar;43(1):28-35. doi: 10.1097/jwh.0000000000000117. PMID 34135723
- [Result] Sanchez-Sanchez F, Ferrer-Casanova C, Ponce-Buj B, Sipan-Sarrion Y, Jurado-Lopez AR, San Martin-Blanco C, Tijeras-Ubeda MJ, Ferrandez Infante A. [Design and validation of the second edition of the Women's Sexual Function Questionnaire, FSM-2]. Semergen. 2020 Jul-Aug;46(5):324-330. doi: 10.1016/j.semerg.2020.01.004. Epub 2020 Mar 18. Spanish. PMID 32197978
- [Result] Sanchez-Sanchez B, Navarro-Brazalez B, Arranz-Martin B, Sanchez-Mendez O, de la Rosa-Diaz I, Torres-Lacomba M. The Female Sexual Function Index: Transculturally Adaptation and Psychometric Validation in Spanish Women. Int J Environ Res Public Health. 2020 Feb 5;17(3):994. doi: 10.3390/ijerph17030994. PMID 32033334
- [Result] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Result] Fernandez-Cuadros ME, Kazlauskas SG, Albaladejo-Florin MJ, Robles-Lopez M, Laborda-Delgado A, de la Cal-Alvarez C, Perez-Moro O. [Effectiveness of multimodal rehabilitation (biofeedback plus capacitive-resistive radiofrequency) on chronic pelvic pain and dyspareunia: prospective study and literature review]. Rehabilitacion (Madr). 2020 Jul-Sep;54(3):154-161. doi: 10.1016/j.rh.2020.02.005. Epub 2020 May 6. Spanish. PMID 32441260
- [Derived] Pla AA, Andreu-Povar A, Fabbi L, Esquirol-Caussa J, Lleberia-Juanos J, Gil-Moreno A, Omana MC. Evaluation of the efficacy of Capacitive Resistive Monopolar Radiofrequency at 448 kHz in the physiotherapeutic treatment of female dyspareunia. Contemp Clin Trials Commun. 2025 Jan 10;44:101433. doi: 10.1016/j.conctc.2025.101433. eCollection 2025 Apr. PMID 39886027